## To explore the potential of UCH-L1 as a novel therapeutic and diagnostic target in heart failure

NCT04999995

August 13, 2024

## RESEARCH CONSENT FORM \_\_\_\_Last 4 SSN: \_\_\_\_Date: Subject Name: Title of Study: Diagnostic potential of UCHL1 in acute decompensated heart failure Local Site Investigator: Phone: Study Sponsor: 1. Introduction and Purpose: We are asking for your participation in a research study conducted at the because you are being admitted to the hospital for shortness of breath. Shortness of breath is a common problem and can have many causes. One of the most common is heart failure. Heart failure is a condition where the heart becomes dysfunctional and is not able to pump blood as effectively as it should. One of the consequences of this is that there is a backup of fluid into the lungs causing a sensation of not being able to breathe well, especially when you exert yourself. The reasons for heart failure are many, including long standing high blood pressure and prior heart attacks. Most conditions that lead to heart failure do so by altering the structure of the heart muscles. One of the processes that leads to this alteration involves impairments in cleaning up of proteins that are not working properly within the heart muscle cells. There is an enzyme called UCHL1 that may prevent the heart muscle cells from properly cleaning up bad proteins when faced with injury. We are interested in seeing if this enzyme UCHL1 can be detected in the blood of patients who present with shortness of breath specifically related to heart failure. The purpose of this study is to determine the ability of blood levels of UCHL1 to help us identify patients who have shortness of breath due to heart failure. 2. **ELIGIBILITY TO PARTICIPATE**: You will be eligible to participate in this study if you are admitted to the hospital for shortness of breath, whether it is related to heart failure or not. 3. **DESCRIPTION OF STUDY PROCEDURES** – There will be NO experimental therapies administered as part of this research trial. We will approach you for enrollment into the study on the day of or the day immediately after your admission to the hospital. If you agree to participate in the study, we will ask you to sign the consent document and we will give you a copy of this document. We will also place a copy in your chart. We will then draw a blood sample and we will also request a urine sample as well. Once we have collected your blood and urine samples, we will conduct a test of how much extra water is in your body. In order to perform this test, you will need to lie down on the hospital bed flat for about 5 minutes. During that time, we will place electrode strips to your skin on your arm and leg. The machine that is recording is recording electrical activity through your skin, very similar to how an EKG machine reads your heart activity. At the end of this recording, we will remove the electrodes and the research activities will be completed for the day.

FORM UCHL1 in HF Consent v8 18JUL2024 10-1086

| | RESEARCH CONSENT FORM (Continuation ) |
|---|---|
| Subject Name: Title of Study: Diagnostic potential Local Site Investigator: Phone: | Date: l of UCHL1 in acute decompensated heart failure |
| hospital (whichever happens first). If yo from the hospital. For all patients with h you have lost about 5% of the weight that marker of heart failure, or you are ready also be recording your lab values, vital stand), urine output, and medications you | test for a total of 5 days or until you are discharged from the ou are here longer than 5 days, we will repeat the test at discharge neart failure, we will collect a second blood and urine sample once at you came to the hospital with, had a 20% decrease in a blood for discharge from the hospital (whichever occurs first). We will igns, weight (standing on a scale, or bed scale if you are unable to u receive during your hospital stay for the same amount of time as |
| For patients who are admitted for shortness vital signs, weight, medications one more collect one more sample of blood and uring a second collection of blood and uring second cations and any lab-work that was decreased as 30 days +/- 14 days from your discharge If there is no follow up set up, we will contain the second category. | oordinate with you the best day and time for a research clinic visit via a check that will be mailed to you (unless you have electronic |

## RESEARCH CONSENT FORM

(Continuation Page  $\underline{3}$  of  $\underline{10}$ )

| Subject Name: | Date: |
|---|---|
| Title of Study: Diagnostic pote<br>Local Site Investigator:<br>Phone: | ential of UCHL1 in acute decompensated heart failure |

| Group | Day of admission/or Day after During hospitalization (2) | | At discharge | | At outpatient<br>follow up (up<br>to 30 days<br>following<br>discharge) | | | |
|---|---|---|---|---|---|---|---|---|
| | HF | NoHF | HF | NoHF | HF | NoHF | HF | NoHF |
| Informed consent | X | X | | | | | | |
| Blood collection | X | X | | | X | X | X | |
| Urine collection | Х | X | | | X | X | X | |
| Recording of<br>medical history,<br>medication history,<br>Past labs | X | X | | | | | | |
| Bioimpedance<br>Measurement<br>(measurement of<br>how much extra<br>water is in your<br>body) | х | Х | Х | | Х | | X | |
| Echocardiogram(1) | | | X | X | | | | |
| Recording of lab<br>work, medications | | | х | Х | Х | Х | х | |

FORM

10-1086 updated Feb 2012

UCHL1 in HF Consent v8 18JUL2024

| | RESEARCH CONSENT FORM (Continuation ) |
|---|---|
| Subject Name: | Date: tial of UCHL1 in acute decompensated heart failure |
| (American Heart Association, 2015) HF: heart failure; NoHF: no heart fail (1) Only for those without a recent echospitalization). (2) During hospitalization we will morprespecified endpoint – which is a perdoctors may order. 4. Risks of Participation: Given that you will be subjected to are minimal. will attempt to make blood draws at the performed for your regular care. This collected. Any additional blood draw the veins; there is also the possibility resulting in lingering discomfort or visindividuals for the blood draw and agalready happening for your regular care. Some people may find extra testing, suncomfortable. We anticipate that the during the assessment. If there is an in | continuous models and record values until you reach a recentage of weight loss or change in value of a blood test your this is primarily an observational study, we anticipate that the risks Most of the data collected will be part of routine clinical care. We he same time as any blood draws that already scheduled to be a way we can just add our tubes to that which is already being as may cause some discomfort due to the insertion of the needle into that during the blood draw we could inadvertently injure the vein as in trying to combine the research blood draw with any that is |

FORM 10-1086 updated Feb 2012

| | RESEARCH CONSENT FORM (Continuation Page <u>5</u> of <u>10</u> ) |
|---|---|
| ubject Name: | Date: |
| Citle of Study: Diagnostic po<br>Local Site Investigator: Phone: | otential of UCHL1 in acute decompensated heart failure |
| substance. Very rarely, some pe<br>will not continue the test for you | cople will develop an allergic reaction to the substance. If that occurs, we |
| the ultrasound probe against the<br>echocardiogram only. In additio<br>echocardiogram may identify ne | provided echocardiogram, there may be discomfort from the pressure of chest. We will try to minimize this by performing a limited on, if a recent echocardiogram is not available, the study provided by problems. This may result in emotional distress for some individuals. It as possible in this situation and notify your healthcare providers care can be provided. |
| We recommend you review these | e risks with your healthcare provider(s). |
| The one exception is those who l | There will likely be no direct benefit to you if you decide to participate. have not had a recent echocardiogram. If you had not had a recent yided by the study, then we may identify a problem that was not known ment if one is available. |
| | nt benefit would be realized for future patients with heart failure. If we as an important marker of heart failure, we may be able to use it in the are patients. |
| <b>6. OTHER TREATMENT AVAILA</b> in this study is to not participate. | BLE, ALTERNATIVES TO PARTICIPATION: The alternative to participation |

UCHL1 in HF Consent v8 18JUL2024

FORM 10-1086 updated Feb 2012

| | RESEARCH CONSENT FORM (Continuation ) |
|---|---|
| Subject Name: | Date: HL1 in acute decompensated heart failure |
| will be paid to you via a mailed check (if an EFT not be required to pay for care received in a payments for medical care and services provided apply to all medical care and services provided by 8. INDEMNITY: The will provide any necess participation in this study. You will be treated for exception, at no cost to you. This also pertains to | Il be reimbursed \$30 for travel time/costs. This amount connection has not been established). Participants will esearch project. Some veterans are required to pay coby. These copayment requirements will continue to that are not part of this study. Is sary medical treatment should you be injured by the injury within this facility, with limited non-veteran participants enrolled in approved exceptions would be situations where this facility would din this case the Medical Center Direct of this remergency treatment in a facility. This |
| 9. VOLUNTARY PARTICIPATION Your participation in the study is voluntary. Refu | y, simply notify . Your decision to participate or withdraw it or future |
| FORM 10-1086 updated Feb 2012 | UCHL1 in HF Consent v8 18JUL2024 |

| | RESEARCH CONSENT FORM (Continuation ) |
|---|---|
| Subject Name: | Date: |
| Local Site Investigator: Phone: | UCHL1 in acute decompensated heart failure |
| confidentially. Your medical information, such answers to the questions on the questionnaires summary of the research findings at profession will be reported as part of the entire group of the presented so that none of your personal information of participation: If, during the part of the study you may be removed recover and you or your family decide aggressive medical therapy, we will result from participation in the research (c) Consequences of self-termination from the removed yourself from the study. Let we will stop all study procedures. Some data and samples already acquired may data and samples removed from the study. It was already acquired may determine the participant of the par | ring work up your data suggests that you no longer qualify to yed from the study. If you are deemed to be too sick to so that it would be in the best interest for you to stop smove you from the study. There are no additional costs to the participant that may h. om the study: There is no consequence to you if you decide |

FORM 10-1086 updated Feb 2012

| | RESEARCH CONSENT FORM (Continuation ) |
|---|---|
| | (Continuation 1 age <u>8</u> of <u>10</u> ) |
| Subject Name: | Date: |
| | potential of UCHL1 in acute decompensated heart failure |
| Local Site Investigator: | |
| Phone: | |
| analysis. This is because The future analyses with The specimens will be site investigator. This research project, us (e) Storage of data after stored in a database the protected and can only has designated as having (f) Future economic potential to future financial (g) ClinicalTrials.gov: A http://www.ClinicalTrinformation that can information that can informatio | In the right to access the data, such as a statistician. Sential of this data: It is not known whether the specimens obtained may all profitable products, but that is always possible. In description of this clinical trial will be available on it is included as summary of the results. In the Web site will include a summary of the results. In the Can See It: Health Authorities (government groups, such as the FDA, inical studies are conducted according to established quality and safety at study information. In the Rights: I have read, and/or I have had read to me all the above. I have all have had them answered. I have been told of the risks or discomforts and I understand that I do not have to take part in the study and that my refusal anyolve no penalty or loss of rights to which I am entitled. I may withdraw |
| FORM 10-1086 updated Feb 201 | UCHL1 in HF Consent v8 18JUL2024 |

| | RESEARCH CONSENT FORM (Continuation ) |
|---|---|
| Local Site Investigator: | |
| Phone: | |
| NEGLIGENCE. IF I AM INJUREI | ED THIS INSTITUTION FROM LIABILITY FOR<br>D IN ANY WAY BY MY PARTICIPATION IN THIS STUDY,<br>IAY OR MAY NOT ALLOW ME TO RECEIVE<br>IJURIES. |
| | e are medical problems or questions, I understand that I can contact ; or emergency assistance during evening hours. If any medical this study, the will provide emergency care. |
| Institutional Review Bo | If I wish to speak with someone o discuss problems, concerns, questions, complaints, obtain |
| WILLINGLY AGREE TO JOIN TH | ESEARCH PARTICIPANT EXPLAINED TO ME AND I IS STUDY. I have had the study explained to me, what it is about will receive a signed and dated copy of this consent form. |
| FORM 10-1086 updated Feb 2012 | UCHL1 in HF Consent v8 18JUL2024 |

| | RESEARCH CO<br>(Continuation Page | ONSENT FORM<br><u>10</u> of <u>10</u> ) |
|---|---|---|
| Subject Name: | | <b>:</b> |
| Title of Study: Diagnostic potentia<br>Local Site Investigator:<br>Phone: | al of UCHL1 in acute decompen | sated heart failure |
| I have been given a chance to ask question to my satisfaction. I agree to participate for my own records. My signature below | e in this study. I have received (or will | receive) a copy of this form |
| Print Name of Participant | Signature of Participant | Date |
| Print Name of Legally Authorized Re Signature of Legally Authorized Repr | | Date |
| Print Name of Person Obtaining Cons | sent Signature of Person Obta | aining Consent Date |
| To be completed by the person obtain Please initial to indicate you have given in Research brochure with the Patient R Additional comments: | the research participant a copy of the V | Volunteering |